CLINICAL TRIAL: NCT00000682
Title: A Randomized, Unblinded Trial of Zidovudine Versus ddC in the Treatment of Patients Status Post PCP Who Received Long-Term Zidovudine Therapy in Protocol ACTG 002
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: ACTG 112; 11087 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Pneumonia, Pneumocystis carinii; Zalcitabine; Acquired Immunodeficiency Syndrome; Zidovudine
MeSH Terms: conditions — HIV Infections; AIDS-Related Opportunistic Infections; Pneumonia, Pneumocystis; Acquired Immunodeficiency Syndrome | interventions — Zidovudine; Zalcitabine

INTERVENTIONS:
Drug: Zidovudine
Drug: Zalcitabine

SUMMARY:
To evaluate the efficacy of AZT versus ddC in terms of survival, antiviral effects, neurological status, and health status in patients post Pneumocystis carinii pneumonia (PCP) who received long-term AZT therapy in ACTG protocol 002 While treatment with AZT has been found to be effective in prolonging survival and reducing the numbers of opportunistic infections in patients with AIDS, during the second year of administration of AZT an acceleration in mortality has been observed. The reasons for this are not known at this time. The study of what may be an AZT-resistant strain of HIV may benefit patients who have been and are still receiving AZT or another drug used in treating HIV ddC. It is hoped that the comparison of the effectiveness of AZT and ddC will benefit in the treatment of these patients.

DETAILED DESCRIPTION:
While treatment with AZT has been found to be effective in prolonging survival and reducing the numbers of opportunistic infections in patients with AIDS, during the second year of administration of AZT an acceleration in mortality has been observed. The reasons for this are not known at this time. The study of what may be an AZT-resistant strain of HIV may benefit patients who have been and are still receiving AZT or another drug used in treating HIV ddC. It is hoped that the comparison of the effectiveness of AZT and ddC will benefit in the treatment of these patients.

Following tests to evaluate their health, patients are chosen at random to receive either AZT or ddC. AZT is given by mouth at the patients' current dose. ddC is given by mouth every 8 hours. Treatment continues for up to 12 months. Patients are required to visit the clinic every 2 weeks up to week 12 and then once a month. Blood samples are taken to monitor the safety and effectiveness of treatment.

ELIGIBILITY:
Inclusion Criteria

Required:

* Prior zidovudine (AZT) therapy for 9 months.

Concurrent Medication:

Allowed:

* Chemoprophylaxis for Pneumocystis carinii pneumonia (PCP) with aerosolized pentamidine of 300 mg every 4 weeks through the Respirgard II nebulizer.
* Maintenance treatment with pyrimethamine, sulfadiazine, amphotericin, fluconazole, ketoconazole, acyclovir, or inhaled pentamidine for subjects who have recovered from toxoplasmosis, cryptococcosis, candidiasis, herpes infection, or PCP.
* Dapsone for PCP.
* Pyrimethamine-sulfadoxine for toxoplasmosis.
* Ganciclovir (DHPG) for maintenance only for cytomegalovirus (CMV) retinitis.
* Note: Any approved medications can be used to treat an opportunistic infection. All concurrent medications should be kept to a minimum and recorded.

Patients must be positive for HIV by ELISA test and must have been receiving zidovudine (AZT) therapy for at least 9 months and have received AZT within 90 days prior to entry into the study.

Patients may be transfusion dependent as long as no more than 3 units of blood are needed in a 21-day period and the hemoglobin does not fall below 6.4 g/dl on two consecutive occasions despite the transfusions.

Exclusion Criteria

Concurrent Medication:

Excluded:

* Antiretroviral study medications other than zidovudine (AZT) and biologic response modifiers.
* Corticosteroids and chronic aspirin.
* Cimetidine.
* Flurazepam.
* Indomethacin.
* Ranitidine.
* Probenecid.
* Other experimental medications.

Patients will be excluded from the study for the following reasons:

* Removal from zidovudine (AZT) during treatment on ACTG protocol 002 for recurrent grade 4 toxicity.
* Removal from prior dideoxycytidine (ddC) therapy for peripheral neuropathy = or > grade 3.
* Visceral or extensive Kaposi's sarcoma requiring therapy or another malignancy requiring therapy.
* Toxicity grades according to NIAID Recommendations for Grading Acute and Subacute Toxic Effects (Adults).

Prior Medication:

Excluded:

* Antiretroviral study medications other than zidovudine (AZT) and biologic response modifiers.
* Patients may not have visceral or extensive Kaposi's sarcoma requiring therapy or another malignancy requiring therapy.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120
Dates: Study Completion 1992-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fischl M, Study Chair; Richman D, Study Chair; Murray H, Study Chair
Locations (5):
- United States (5):
  - USC CRS, Los Angeles, California
  - Ucsd, Avrc Crs, San Diego, California
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Pitt CRS, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Henry K, Tierney C, Kahn J, Balfour H, Jiang Q, Kmack A, Fischl M. A randomized, double-blind, placebo-controlled study comparing combination nucleoside and triple therapy for the treatment of advanced HIV disease (CD4 less than or equal to 50/mm(3)). Conf Retroviruses Opportunistic Infect. 1997 Jan 22-26;4th:207 (abstract no LB6)
- [Background] Skowron G, Bozzette SA, Lim L, Pettinelli CB, Schaumburg HH, Arezzo J, Fischl MA, Powderly WG, Gocke DJ, Richman DD, Pottage JC, Antoniskis D, McKinley GF, Hyslop NE, Ray G, Simon G, Reed N, LoFaro ML, Uttamchandani RB, Gelb LD, Sperber SJ, Murphy RL, Leedom JM, Grieco MH, Zachary J, Hirsch MS, Spector SA, Bigley J, Soo W, Merigan TC. Alternating and intermittent regimens of zidovudine and dideoxycytidine in patients with AIDS or AIDS-related complex. Ann Intern Med. 1993 Mar 1;118(5):321-30. doi: 10.7326/0003-4819-118-5-199303010-00001. PMID 8094279